CLINICAL TRIAL: NCT04427969
Title: The Effect of Early Prone Position on Prognosis in Acute Respiratory Failure Due to Coronavirus Disease 2019 Pneumonia
Brief Title: Early Prone Position on Coronavirus Disease 2019 Pneumonia
Acronym: Prone Position
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mustafa Altınay, spercialist medical doctor, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: pp34
Record Dates: First submitted 2020-06-06; First posted 2020-06-11 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Coronavirus Infection; Acute Respiratory Failure
Keywords: coronavirus disease 2019; prone position
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Prone Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EPP: patients who applied early awake prone position for treatment with conventional oxygen supply
  Interventions: Behavioral: prone position
- non-EPP: patient who only get conventional oxygen therapy as respiratory supply

INTERVENTIONS:
Behavioral: prone position — to lay in prone position at least 12 hour in a day at ICU
  Groups: EPP

SUMMARY:
the purpose of this study to evaluate the effect of early awake PP (prone position)application on oxygenation and intubation requirement in patients with acute respiratory failure due to coronavirus disease 2019 pneumonia.

DETAILED DESCRIPTION:
The first group (early prone position-EPP) created for our study was composed of patients who received PP at least 12 hours early (with the first 48 hours) with the oxygen support of the reservoir mask, and the second group (non-EPP ) patients who received oxygen with the reservoir mask but could not be applied early PP due to the patient's incompatibility or rejection.

Conventional oxygen therapy applied to all patients was given with a reservoir mask, aiming at oxygen saturation 93% and above, at a flow rate of 6-15 L / min.

Despite all the treatments, the patients who have a follow-up with a respiratory acidosis , oxygen saturation value below 93%, applied non invasive mechanical ventilation, in case of insufficient patient intubated and have invasive mechanical ventilation. In patients who had regression of glasgow coma scale during follow-up, orotracheal intubation was performed and invasive mechanical ventilation was performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who developed acute respiratory failure due to coronavirus disease 2019 pneumonia
* received conventional oxygen therapy with reservoir mask oxygen at the stage of admission to the intensive care unit
* older than 18 years old

Exclusion Criteria:

* patients with respiratory acidosis,
* partial oxygen pressure/fraction of inspired oxygen ratio below 150,
* Glasgow Coma Score (GKS) below 12 points,
* hemodynamic instability,
* primary pulmonary pathologies other than pneumonia (lung cancer, cardiopulmonary edema, carcinogen syndrome, etc.)
* patients who underwent non-invasive mechanical ventilation(NIMV) or intubated from admission to intensive care,
* those who underwent self prone position under 12 hours were not included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data of patients over 18 years old who were followed up and treated in the intensive care unit due to acute respiratory failure due to coronavirus disease 2019 pneumonia were retrospectively reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-06-25 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
intensive care unit stay | up to 28 days
  the duration of icu stay day
short term mortality | up to 28 days
  mortality percent

SECONDARY OUTCOMES:
blood gases | up to 24 hours
  partial oxygen pressure: mmhg , partial carbondiocsit pressure mmhg

CONTACTS AND LOCATIONS:
Overall Officials: ayse surhan cinar, Study Chair — chief of anesthesia department
Locations (1):
- Sisli Etfal Research and Training Hospital, Istanbul, Marmara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Result] Guerin C, Reignier J, Richard JC, Beuret P, Gacouin A, Boulain T, Mercier E, Badet M, Mercat A, Baudin O, Clavel M, Chatellier D, Jaber S, Rosselli S, Mancebo J, Sirodot M, Hilbert G, Bengler C, Richecoeur J, Gainnier M, Bayle F, Bourdin G, Leray V, Girard R, Baboi L, Ayzac L; PROSEVA Study Group. Prone positioning in severe acute respiratory distress syndrome. N Engl J Med. 2013 Jun 6;368(23):2159-68. doi: 10.1056/NEJMoa1214103. Epub 2013 May 20. PMID 23688302
- [Result] Kallet RH. A Comprehensive Review of Prone Position in ARDS. Respir Care. 2015 Nov;60(11):1660-87. doi: 10.4187/respcare.04271. PMID 26493592
- [Result] Munshi L, Del Sorbo L, Adhikari NKJ, Hodgson CL, Wunsch H, Meade MO, Uleryk E, Mancebo J, Pesenti A, Ranieri VM, Fan E. Prone Position for Acute Respiratory Distress Syndrome. A Systematic Review and Meta-Analysis. Ann Am Thorac Soc. 2017 Oct;14(Supplement_4):S280-S288. doi: 10.1513/AnnalsATS.201704-343OT. PMID 29068269

DOCUMENTS (2):
  • Study Protocol (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT04427969/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT04427969/SAP_001.pdf